CLINICAL TRIAL: NCT05380908
Title: The Fifth Affiliated Hospital of Sun Yat-sen University
Brief Title: Brain Metabolic Network of PET in Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: K059(2021-059)
Record Dates: First submitted 2022-05-13; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Advanced Non-small-cell Lung Cancer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with untreated non-small cell lung cancer
  Interventions: Other: None of any intervention
- Patients with non-small cell lung cancer after chemotherapy
- Normal controls
  Interventions: Other: None of any intervention

INTERVENTIONS:
Other: None of any intervention — The patients did not have any intervention.
  Groups: Normal controls; Patients with untreated non-small cell lung cancer

SUMMARY:
This study is a retrospective study, screening patients with systemic PET / CT scan in our department, enrolling the ones who meet the criteria, collect their information and resting state brain PET images.Then make the brain metabolic network analysis and statistical analysis to explore the PET brain metabolic network of non-small cell lung cancer patients and the effect of chemotherapy drugs on brain metabolic network in patients with advanced lung cancer.

DETAILED DESCRIPTION:
1. Enroll Participants
2. Collect PET/CT Images
3. Images Analysis
4. Statistical Analysis

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced non-small cell lung cancer without any treatment and pathological confirmed non-small cell lung cancer.

Exclusion Criteria:

* Brain tumors (primary or metastasis), previous surgery, radiotherapy, chemotherapy, stroke, head trauma, psychiatric history (insomnia, depression, mania, schizophrenia and other psychiatric disorders), or history of drug dependence (e. g. sedatives, sleeping pills or sedatives)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with pathological confirmed non-small cell lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Death | 1-5 years

CONTACTS AND LOCATIONS:
Locations (1):
- PET/CT, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: No